CLINICAL TRIAL: NCT05139563
Title: South African Male User Research on Acceptability of Implants and Injections
Acronym: SAMURAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 00021779; 00021820 (Other: RTI International)
Record Dates: First submitted 2021-11-04; First posted 2021-12-01 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Acceptability
MeSH Terms: interventions — soybean oil, phospholipid emulsion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo injection (Sham Comparator): This group will first receive 3 mL intramuscular injections of a 20% fat emulsion (Intralipid 20%) every 2 months for 6 months.
  Interventions: Other: Placebo injection: Intralipid 20% fat emulsion; Other: Placebo implant
- Placebo implant (Experimental): This group will first receive a single-use subdermal implant in the inner side of the upper arm for a duration of 6 months before removal.
  Interventions: Other: Placebo injection: Intralipid 20% fat emulsion; Other: Placebo implant

INTERVENTIONS:
Other: Placebo injection: Intralipid 20% fat emulsion — placebo intralipid 20% intramuscular (IM) injection
Other: Placebo implant — placebo subdermal implant rod

SUMMARY:
The overall aims of SAMURAI (South African Male User Research on Acceptability of Implants and Injections) are to assess acceptability of, and preferences for, novel long-acting pre-exposure prophylaxis (LA-PrEP) delivery formulation use among key end-users: heterosexual men and men-who-have-sex-with-men (MSM) in South Africa, a country most impacted by human immunodeficiency virus (HIV) incidence and prevalence. Early involvement of men in product development is an important opportunity to measure and address product acceptability and factors that may influence adherence and to foster male ownership of novel HIV prevention delivery modalities.

DETAILED DESCRIPTION:
Long-acting (LA) pre-exposure prophylaxis (PrEP) offers a promising alternative to existing HIV prevention methods. Research to assess end-user acceptability and actual experiences of novel delivery formulations has neglected, however, to include male perspectives, despite these products being appropriate for use by both men and women. This research aims to assess acceptability of and preferences for novel LA PrEP delivery formulation use among key end users: heterosexual men and men who have sex with men (MSM) in South Africa. Early involvement of men in product development is an important opportunity to measure and address product acceptability and foster male ownership of novel strategies, thereby enhancing potential effectiveness and impact, and broadening male engagement in HIV prevention.

LA PrEP delivered by implant or injection addresses user preferences for simplicity, discretion, and longer dose duration. Currently, there are several PrEP implants in preclinical development and a few injectable formulations in early human phase trials. Biomedical strategies have two core components: the active pharmaceutical ingredient and the delivery mechanism; both of which contribute to acceptability and successful use of products. Research to assess acceptability of placebo use of LA PrEP delivery forms among end users provides insight that may apply to the many products under development. The contraceptive field provides substantial information about potential acceptability and use of LA delivery methods among women in sub-Saharan Africa (SSA). However, there is a gap in knowledge regarding acceptability of implant and injectable dosing platforms among men, particularly in SSA.

The investigators propose a four-year study to comparatively examine acceptability and preferences of placebo implants and injectables using a crossover-designed mixed methods study among heterosexual men and MSM in Johannesburg and Cape Town, South Africa. The investigators hypothesize that men will find implant use acceptable as a delivery form and no less acceptable than intramuscular injections. First, formative qualitative research with men (n=40) will be conducted to assess knowledge and experiences and inform messages and materials for our Aim 2 and 3 work. Subsequently, a clinical crossover study will be conducted, in which men (n=200) will wear placebo implants for 6 months and have three bimonthly injections in a randomized sequence. Preferences for these delivery forms and product attributes of these LA methods, oral PrEP, and condoms will then be measured using a discrete choice experiment survey.

ELIGIBILITY:
Inclusion Criteria:

1. Being cis-gender male per self-identification
2. Aged 18-35 years
3. In good physical health, as determined by the site investigator or designee based on clinical history
4. Willing and able to comply with study procedures and attend follow-up visits over 1 year
5. Fluent in English, Xhosa, or Zulu
6. Sexually active, defined by receptive or insertive anal or vaginal intercourse at least once a month in the past 3 months
7. Able and willing to comply with all study procedural requirements
8. Able and willing to provide informed consent
9. Intention to stay within study catchment area for study duration and willingness to give adequate locator information
10. At Screening and Enrollment, states a willingness to refrain from participation in other research studies involving drugs, vaccines, or medical devices during study participation. Participation in other behavioral studies is subject to Investigator discretion.

Exclusion Criteria:

1. Known or suspected allergy to study product components (active or placebo), including egg or soy products (egg and soy products are contained in Intralipid).
2. At Screening or Enrollment, has a positive HIV test.
3. Diagnosed or suspected sexually transmitted infection (STI) requiring treatment at Enrollment such as gonorrhea (GC), chlamydia, trichomonas, and/or syphilis. Enrollment will be considered after treatment of STIs.

   Note: Genital warts requiring treatment and frequent recurrence of herpes simplex virus (HSV) are considered exclusionary; however, infrequent HSV outbreaks are not. Genital warts requiring treatment are defined as those that cause undue burden or discomfort to the participant, including bulky size, unacceptable appearance, or physical discomfort.
4. As determined by the Investigator/designee, any current or historical physical or mental health condition that the site investigator or designee determines should exclude participation (for example, injection drug use within the past year).
5. Has any other condition that, in the opinion of the Investigator/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
6. At Enrollment, participant reports current or recent (30 days or less prior to enrollment) participation in any research study involving drugs, vaccines, or medical devices. Allowance for co-enrollment in other types of studies is indicated below.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender men
Enrollment: 184 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Product initial attitudes rating (4-point Likert scale) | Baseline
  Assessment of participants' attitudes towards placebo long-acting (LA) PrEP study product physical attributes, expected ease of use, delivery method, and expected physical discomfort
Product satisfaction rating (4-point Likert scale) | Month 6
  Assessment of participants' satisfaction with placebo long-acting (LA) PrEP study product physical attributes, ease of use, delivery method, and physical discomfort
Product satisfaction rating (4-point Likert scale) | Month 12
  Assessment of participants' satisfaction with placebo long-acting (LA) PrEP study product physical attributes, ease of use, delivery method, and physical discomfort
Adherence to study product regimen | throughout study completion, average 1 year
  Documentation of initiation and sustained use of placebo LA-PrEP study product

SECONDARY OUTCOMES:
Assessment of Adverse Events (AEs) for study product delivery methods | throughout study completion, average 1 year
  Number, relatedness, and severity of reported AEs and serious adverse events
Assessment of Social Harms | throughout study completion, average 1 year
  Number and severity of Social Harms (i.e., non-medical adverse consequences of participation such as discrimination, stigma, abuse, etc.) reported by participants
Preference comparison for PrEP Delivery method | Month 12
  Self-comparison of participants' stated preferences of currently available and possible PrEP delivery methods [i.e., discrete choice experiment (DCE)] implemented at the exit clinical study visit. Investigators will assess preferences for implants as compared with injections; as well as preferences for product-specific attributes of each approach.
Burden of placebo product-specific pain | throughout study completion, average 1 year
  Assessed by participant self-reported rating of physical pain from placebo product administration using a 10-point visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Montgomery, PhD, Principal Investigator — RTI International
Locations (2):
- South Africa (2):
  - Desmond Tutu Health Foundation, Philippi Village, Cape Town
  - Wits RHI, Johannesburg

IPD SHARING:
Plan to Share IPD: Undecided